CLINICAL TRIAL: NCT01498302
Title: Interlaboratory Comparability Study of Residual Disease in Acute Myelogenous Leukemia
Brief Title: Comparison of Laboratory Test Results of Minimal-Residual Disease in Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B5; COG-AAML12B5 (Other: Children's Oncology Group); AAML12B5 (Other: Children's Oncology Group); NCI-2012-00098 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-22; First posted 2011-12-23 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Bone marrow and/or peripheral blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis
Other: flow cytometry

SUMMARY:
RATIONALE: Diagnostic procedures that find residual disease may help predict if the disease will come back in patients diagnosed with acute myeloid leukemia.

PURPOSE: This research trial studies the comparison of laboratory test results for minimal residual disease in samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To promote harmonization between Cooperative Group Reference Laboratories conducting minimal-residual disease (MRD) evaluation of acute myeloid leukemia by flow cytometry.

OUTLINE: Archived bone marrow and blood samples, distributed to the Eastern Cooperative Oncology Group, Southwest Oncology Group, and Cancer and Leukemia Group B laboratories, are analyzed for leukemia-associated immunophenotype (LAIP) assays and minimal residual disease studies by flow cytometry. Results are then provided to the National Cancer Institute for assessment and comparability of test results.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Non-identified cryopreserved samples of bone marrow and/or peripheral blood from patients with acute myeloid leukemia (AML) from the Children Oncology Group (COG) studies

  * Baseline/diagnostic AML samples
  * Samples collected after initial treatment and representing varying levels of residual blast counts

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute myeloid leukemia (AML) enrolled on Children's Oncology Group (COG) studies.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Degree of concordance in the MRD assay results between laboratories

CONTACTS AND LOCATIONS:
Overall Officials: J. Milburn Jessup, MD, Principal Investigator — National Cancer Institute (NCI)